CLINICAL TRIAL: NCT02844933
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study to Assess the Efficacy, Safety, and Tolerability of Cannabidiol Oral Solution for the Treatment of Patients With Prader-Willi Syndrome
Brief Title: Cannabidiol Oral Solution for the Treatment of Patients With Prader-Willi Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insys Therapeutics filed Chapter 11 and terminated all studies.
Sponsor: Radius Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INS011-16-085
Record Dates: First submitted 2016-07-22; First posted 2016-07-26 (Estimated); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (Experimental): Cannabidiol oral solution (40 milligram/kilogram/day [40 mg/kg/day]) divided into two daily doses with a standard meal
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator): Matching placebo solution divided into two daily doses with a standard meal
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — Oral solution
  Arms: Cannabidiol
Drug: Placebo — Matching oral solution
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the efficacy of cannabidiol oral solution on hyperphagia-related behavior in patients with Prader-Willi Syndrome (PWS). The secondary objectives of this study are to assess the efficacy, safety and tolerability, impact on quality of life, and impact on physical activity of cannabidiol oral solution in patients with PWS.

ELIGIBILITY:
Inclusion Criteria:

* Participant and/or parent(s)/caregiver(s) fully comprehend the informed consent form and assent form, understand all study procedures, and can communicate satisfactorily with the investigator and study coordinator, in accordance with applicable laws, regulations, and local requirements.
* Participants with a genetically confirmed diagnosis of Prader-Willi Syndrome using standard deoxyribonucleic acid methylation test or fluorescent in situ hybridization. Documentation of genetically confirmed diagnosis of Prader-Willi Syndrome is acceptable.
* A score of ≥10 on the Hyperphagia Questionnaire for Clinical Trials (HQ-CT).
* A caregiver is available to complete the HQ-CT.
* If female, is either not of childbearing potential (defined as premenarchal or surgically sterile [bilateral tubal ligation, bilateral oophorectomy, or hysterectomy]) or practicing one of the following medically acceptable methods of birth control:

  1. Hormonal methods such as oral, implantable, injectable, vaginal ring, or transdermal contraceptives for a minimum of 1 full cycle (based on the participant's usual menstrual cycle period) before study drug administration.
  2. Total abstinence from sexual intercourse since the last menses before study drug administration.
  3. Intrauterine device.
  4. Double-barrier method (condoms, sponge, or diaphragm with spermicidal jellies or cream).
* Adequate renal function, defined as serum creatinine ≤ 1.5*upper limit of normal (ULN) and urine protein/creatinine ratio ≤0.4. The Investigator may deem the participant eligible if he or she judges the laboratory values to be not clinically significant.
* Adequate hepatic function, defined as total bilirubin ≤ 1.5*ULN and aspartate aminotransferase and alanine aminotransferase levels ≤ 3*ULN.
* Growth hormone treatment will be permitted if doses have been stable for at least 1 month prior to screening.
* Psychotropic treatment will be permitted and should be stable at least 6 weeks prior to screening.
* Any other treatment including thyroid hormones should be stable for at least 6 weeks prior to screening.

Exclusion Criteria:

* Known use of cannabis or cannabinoid-containing products for 4 weeks prior to baseline.
* History of chronic liver diseases, such as cirrhosis or chronic hepatitis due to any cause, or suspected alcohol abuse.
* Use of weight loss agents or drugs known to affect appetite (including glucagon-like peptide-1 [GLP-1] analogs) within 2 months prior to screening.
* Uncontrolled Type I and Type II diabetes.
* Currently taking concomitant medication that are strong-moderate inhibitors/inducers/sensitive substrates with a narrow therapeutic index for CYP2C19 or CYP3A.
* Co-morbid condition or disease (such as respiratory disease, heart disease, or psychiatric disorder) diagnosed less than 1 month prior to screening.
* History or presence of gastrointestinal or any other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs as determined by the Investigator.
* Participants who have participated in any other trials involving an investigational product or device within 30 days of screening or longer as required by local regulations.
* Clinically significant abnormalities on electrocardiogram at screening or other evidence of heart disease as determined by the Investigator.
* Has screening systolic blood pressure ≥160 millimeters of mercury (mmHg) and diastolic blood pressure >100 mm Hg (may be repeated 1 additional time after 5 minutes rest to verify). Participants with hypertensive levels lower than those specified may be excluded at the Investigator's discretion if deemed to be in the best interest of the participant.
* Currently taking felbamate.
* Uncontrolled sleep apnea.
* Pregnant or lactating female.
* History of hypersensitivity to drugs with a similar chemical structure or class as cannabidiol.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Participant judged by the investigator or sponsor (or designee) as unable to comply with the treatment protocol, including appropriate supportive care, follow-up and research tests.
* Positive drug screen, including tetrahydrocannabinol, at time of screening.
* Creatinine clearance test of < 30 milliliters/minute (mL/min).

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elkashef, MD, Study Director — INSYS Therapeutics Inc
Locations (7):
- United States (7):
  - University of Arizona, Tucson, Arizona
  - Rady Children's, UC San Diego, San Diego, California
  - University of Iowa, Iowa City, Iowa
  - The University of Kansas , Medical Center, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - The University of Oklahoma Health Sciences Center, Tulsa, Oklahoma
  - Institute for Research and Innovation | MultiCare Health System, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in the United States from 09 May 2018 and 31 July 2019.
Pre-assignment Details: Approximately 66 participants aged 8 to 17 years, inclusive, with a genetically confirmed diagnosis of Prader-Willi Syndrome were planned to be enrolled in the study. The previous Sponsor prematurely terminated the study prior to reaching the planned enrollment. Therefore, only 7 participants participated in the study.
Groups:
- Cannabidiol: Participants received cannabidiol oral solution of 40 milligram/kilogram/day (mg/kg/day) divided into two daily doses with a standard meal.
- Placebo: Participants received a matching placebo solution divided into two daily doses with a standard meal.
Period: Overall Study
Arm/Group | Cannabidiol | Placebo
Started | 4 | 3
Received at Least 1 Dose of Study Drug | 4 | 3
Completed | 1 | 1
Not Completed | 3 | 2
Not completed — Discontinued due to premature termination of study | 3 | 2

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled and received at least 1 dose of study drug.
Groups:
- Cannabidiol: Participants received cannabidiol oral solution (40 mg/kg/day) divided into two daily doses with a standard meal.
- Placebo: Participants received matching placebo solution divided into two daily doses with a standard meal.
- Total: Total of all reporting groups
Arm/Group | Cannabidiol | Placebo | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Mean (Full Range); unit: years] | 13.5 [10 to 15] | 11.67 [8 to 15] | 12.7 [8 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Baseline in Total Body Weight [Median (Full Range); unit: kg] — Total body weight refers to the participants weight throughout the study.
  kg | 88.35 [47.9 to 112.4] | 56.7 [45.5 to 109.7] | 72.50 [45.5 to 112.4]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hyperphagia Behavior as Measured by the Hyperphagia Questionnaire for Clinical Trials (HQ-CT)
Description: The HQ-CT measures hyperphagia by Prader-Willi syndrome (PWS)-specialized clinicians. The HQ-CT generates a score ranging from 0 to 36, where a higher score represents more severe abnormal food related behaviors.
  The change from baseline was calculated from two time points as the value at the later time point minus the value at the earlier time point: value at Week 13 minus value at Baseline.
Time Frame: Baseline, Week 13
Population: All participants who received at least 1 dose of study drug
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Cannabidiol | Placebo
Number analyzed (Participants) | 4 | 3
score on a scale
  Baseline | 23 [10 to 25] | 22 [18 to 26]
  Week 13 | 14 [7 to 20] | 16 [10 to 28]
  Change from Baseline at Week 13 | -4.5 [-14 to -3] | -2 [-12 to 2]

2. Secondary Outcome: Change From Baseline In Total Body Weight
Description: Total body weight refers to participants' weight throughout the study. The change from baseline was calculated from two time points as the value at the later time point minus the value at the earlier time point: value at Week 13 minus value at Baseline.
Time Frame: Baseline, Week 13
Population: All participants who received at least 1 dose of study drug
Measure: Median (Full Range); unit: kg
Arm/Group | Cannabidiol | Placebo
Number analyzed (Participants) | 4 | 3
kg
  Baseline | 88.35 [47.9 to 112.4] | 56.7 [45.5 to 109.7]
  Week 13 | 87.6 [47.4 to 110.8] | 59.5 [46.8 to 109.4]
  Change From Baseline at Week 13 | -1.05 [-1.6 to 0.1] | 1.3 [-0.3 to 1.3]

3. Secondary Outcome: Responder Rate From Baseline Through Study Completion
Description: A responder was defined as having a 6 or more points decrease in HQ-CT score.
Time Frame: Baseline up to Week 13
Population: All participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol | Placebo
Number analyzed (Participants) | 4 | 3
Participants
  Yes | 1 | 1
  No | 3 | 2

4. Secondary Outcome: Change In Patient Global Impression Of Change (PGI-C) Questionnaire
Description: The change in PGI-C scores at Week 3, Week 9, and Week 13 of the participant are evaluated.
Time Frame: Week 3, Week 13
Population: Due to early study termination, data was not collected for analysis of this outcome measure.
Arm/Group | Cannabidiol | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline In The Three Factor Eating Questionnaire - 18-item Version (TFEQ-R18)
Description: The change from baseline to Week 13 of the participant's TFEQ-R18 score is evaluated.
Time Frame: Baseline, Week 13
Population: Due to early study termination, data was not collected for analysis of this outcome measure.
Arm/Group | Cannabidiol | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline In Quality Of Life [Patient-Reported Outcomes Measurement Information System (PROMIS) Life Satisfaction And Positive Affect Questionnaires]
Description: The change from baseline to Week 13 of the participant's quality of life (PROMIS life satisfaction and positive affect questionnaire) score is evaluated.
Time Frame: Baseline, Week 13
Population: Due to early study termination, data was not collected for analysis of this outcome measure.
Arm/Group | Cannabidiol | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline In Physical Activity (PROMIS Physical Activity And Fatigue Questionnaires)
Description: The change from baseline to Week 13 of the participant's physical activity (PROMIS physical activity and fatigue questionnaires) score is evaluated.
Time Frame: Baseline, Week 13
Population: Due to early study termination, data was not collected for analysis of this outcome measure.
Arm/Group | Cannabidiol | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 13
Description: Safety population included all participants who received at least 1 dose of study medication.
Arm/Group | Cannabidiol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 4/4 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cannabidiol (N=4) | Placebo (N=3)
Diarrhea (Gastrointestinal disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Abdominal cramping (Gastrointestinal disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Seizure (Nervous system disorders) | 0 | 1
Impetigo (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Ear infection (Ear and labyrinth disorders) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0

LIMITATIONS AND CAVEATS:
This study was prematurely terminated by the previous Sponsor (Insys Therapeutics Inc.). Only 7 participants were enrolled, and the planned number of participants was not achieved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/33/NCT02844933/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/33/NCT02844933/SAP_001.pdf